CLINICAL TRIAL: NCT05049980
Title: Evaluation of the Efficacy, Tolerance of the Treatment, and Patient Satisfaction During the Management of an Arrested Pregnancy in the First Trimester According to the New Toulouse University Hospital Protocol
Brief Title: Patient Satisfaction With the Management of a Stopped Pregnancy in the First Trimester
Acronym: MYFEFACY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0328
Record Dates: First submitted 2021-08-26; First posted 2021-09-20 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Loss, Early
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical treatment (Experimental): Patients choosing medical treatment with Mifégyne® and MisoOne®
  Interventions: Drug: Medical treatment with Mifégyne® and MisoOne®
- Surgical treatment (Active Comparator): Patients choosing surgical treatment by endo-uterine aspiration.
  Interventions: Procedure: Endo-uterine aspiration

INTERVENTIONS:
Drug: Medical treatment with Mifégyne® and MisoOne® — When participants arrive for their uterine emptiness check-up, 12 days after treatment, patients will be asked to drop off the study questionnaire the same day in a box provided for this purpose in the department.
  Arms: Medical treatment
Procedure: Endo-uterine aspiration — When patients arrive in hospital on the day of the surgery, participants will be asked to complete a questionnaire at home 1 week after surgery and return it to investigators.
  Arms: Surgical treatment

SUMMARY:
The clinical practice recommendations highlight the fact that the patient's choice concerning the management of her aborted pregnancy in the first trimester should be privileged, after clear and appropriate information on the available treatments, in order to improve his experience and reduce the negative psychological symptoms that can generate an alteration in the quality of life, in the aftermath of the loss of pregnancy.

The present study will describe the efficacy, satisfaction and tolerance of patients benefiting from medical treatment with Mifégyne® and MisoOne® versus those benefiting from surgical treatment by endo-uterine aspiration for the management of a pregnancy stopped during the first trimester at the Toulouse University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient presenting to the gynecological emergency department of the Paule de Viguier Hospital in Toulouse for whom a diagnosis of an arrested pregnancy in the first trimester is made
* Whose cranio-caudal length of the embryo measured by ultrasound is less than 25 mm or having a clear egg
* Having agreed to the study (written or verbal) after clear and fair information
* Who understands and reads French

Exclusion Criteria:

* Medical contraindication to treatment with Mifégyne® or MisoOne®
* Hemodynamically unstable patient requiring urgent surgical treatment.
* Protected adult patient (guardianship, curatorship, safeguard of justice)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Inclusion day (day 0)
Patient satisfaction | Inclusion day (day 0)
  Completing the satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mickael ALLOUCHE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Mickael ALLOUCHE, Toulouse, France

IPD SHARING:
Plan to Share IPD: No